CLINICAL TRIAL: NCT02118324
Title: The Effect of a Home-based Fitness Intervention on Cardiometabolic Risk Profile in Acute Lymphoblastic Leukemia (ALL) Patients
Brief Title: Exergaming Intervention in ALL Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013NTLS119
Record Dates: First submitted 2014-03-26; First posted 2014-04-21 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; ALL; fitness intervention
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise treatment (Experimental): Participants will be instructed to use the exergaming program at home for 30 mins, 3-5 times per week.
  Interventions: Behavioral: Exergaming Program
- Control group (No Intervention): No intervention is provided.

INTERVENTIONS:
Behavioral: Exergaming Program — Participants will exercise through exergaming play.
  Arms: Exercise treatment

SUMMARY:
This is a pilot feasibility study to collect preliminary data for a large-scale exergaming intervention in children undergoing maintenance therapy for Acute Lymphoblastic Leukemia (ALL). Patients, ages 5-17 years will be randomized to the intervention or non-intervention control group. The intervention will consist of 30 minute sessions of exergaming 3-5 times a week for 6 months, with weekly assessment of exercise level and phone calls by kinesiology graduate students for safety and compliance. Physical activity at baseline and at the end of study will be assessed using accelerometers. Outcome measures will include: anthropometrics, blood pressure, body composition, visceral fat, vascular function, fasting insulin, fasting glucose, LDL-cholesterol, HDL- cholesterol, triglycerides, functional mobility and endurance, and strength.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility will not be restricted by race or sex
* Pediatric patients with ALL diagnosis, treated at the University of Minnesota Amplatz Children's Hospital or Children's Hospitals and Clinics of Minnesota
* At least 3 months into the maintenance phase, with at least 6 months left of maintenance therapy
* Age 5-17 years at time of study enrollment
* Not smoking
* Currently not involved in a regular (3 times per week) exercise program

Exclusion Criteria:

* Individuals with a physical or mental impairment which would preclude their ability to perform the intervention.
* Bone marrow transplant recipients.
* Any woman currently pregnant will not be eligible, but may participate 3 or more months after the end of her pregnancy if the study is still ongoing
* Due to the intervention being in English, non-English speakers will be excluded

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Average minutes of physical activity per day | 6-months
  The feasibility of an exercise intervention in pediatric ALL patients undergoing maintenance therapy and its effects on markers of cardiometabolic risk. The primary outcome for this pilot study is average minutes and time spent at varying intensity of physical activity per day, as measured by accelerometers.

SECONDARY OUTCOMES:
Average difference of blood pressure | 6 months
  Estimate of the likely effect size (i.e., difference between the groups in average outcome) of blood pressure.
Average difference of body composition | 6 months
  Estimate of the likely effect size (i.e., difference between the groups in average outcome) of body composition.
Average difference in visceral fat | 6 months
  Estimate of the likely effect size (i.e., difference between the groups in average outcome) of visceral fat.
Average difference in triglycerides | 6 months
  Estimate of the likely effect size (i.e., difference between the groups in average outcome) of triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Steinberger, MD, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Amplatz Children's Hospital, Minneapolis, Minnesota, United States